CLINICAL TRIAL: NCT05151367
Title: SEARCH: Short Message Service (SMS) Electronic Adolescent Reminders for Completion of HPV Vaccination - Uganda: Pilot
Brief Title: SMS HPV Vaccine Reminders
Acronym: SEARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Makerere University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa Stockwell, Associate Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AAAT1572; 1R21CA253604-01 (NIH)
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Human Papillomavirus Vaccination
Keywords: Human papillomavirus; Vaccination; Text message; SMS; mHealth; Reminder; Uganda

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text message reminders (Experimental): Text message reminders
  Interventions: Behavioral: Text message reminder
- Usual Care (No Intervention): No reminders

INTERVENTIONS:
Behavioral: Text message reminder — Receipt of text messages notifying when the next HPV vaccine dose is due (either first or second)
  Arms: Text message reminders

SUMMARY:
This study will take place at health centres and their affiliated schools and community immunization centers overseen by the Kampala Capital City Authority (KCCA) as well as at the Makerere/Mulago/Columbia Adolescent Health Clinic, also in Kampala. While text messages can be used in populations with low literacy, families can opt to receive automated phone call reminders instead. The investigators will pilot assess the impact of vaccine reminders on human papillomavirus (HPV) vaccination. Caregivers of preteens/adolescents will be randomized and stratified by site, language and HPV vaccine dose needed (initiation vs. completion). As this is a feasibility trial, the investigators expect to measure effect size but not necessarily achieve statistical significance.

DETAILED DESCRIPTION:
Cervical cancer is the leading female cancer in Uganda. Many women are diagnosed with late-stage disease, and 80% of women die within 5 years of diagnosis, making primary prevention critical. HPV is the principal cause of cervical cancer, making vaccination the single most important primary preventive measure. The national HPV vaccination program in Uganda began in November 2015 and focuses solely on preteen/adolescent girls. Two strategies have been adopted for the multi-dose series: 1) school-based and 2) community-based. However, in Kampala, only 29% of girls receive both needed doses. Reasons for undervaccination include school absenteeism on special vaccination days for those receiving vaccination as part of a school program, failing to remember to come to a health facility for a needed dose for those being vaccinated in the community, and lack of knowledge regarding HPV and the vaccines including vaccine misperceptions. While research regarding the use of text message vaccine reminders is strong in the U.S., their use has not yet been demonstrated in a preteen/adolescent population in Sub-Saharan Africa and other low and middle income countries (LMICs). According to the World Bank, currently 89.9% of urban households in Uganda have a cell phone.

ELIGIBILITY:
Inclusion Criteria:

* Be a parenting adult of an adolescent girl aged 10-14 years
* Reside in Kampala and/or the surrounding districts
* Speak English or Luganda
* Have a cell phone with text messaging capability
* Must have ability to consent

Exclusion Criteria:

* Parenting adult speaks other language than English or Luganda only
* Parenting adult already enrolled in the study for another child
* Participation in pretesting activities

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S. Stockwell, MD, MPH, Principal Investigator — Columbia University
Locations (2):
- Columbia University Irving Medical Center, New York, New York, United States
- Makerere University/Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kitaka SB, Rujumba J, Zalwango SK, Pfeffer B, Kizza L, Nattimba JP, Stephens AB, Nabukeera-Barungi N, Wynn CS, Babirye JN, Mukisa J, Mupere E, Stockwell MS. SEARCH Study: Text Messages and Automated Phone Reminders for HPV Vaccination in Uganda: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 May 5;13:e63527. doi: 10.2196/63527. PMID 40324213

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Message Reminders | Usual Care
Started | 78 | 76
Completed | 78 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Message Reminders | Usual Care | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Customized [Count of Participants; unit: Participants]
  10 years | 15 | 17 | 32
  11 years | 20 | 18 | 38
  12 years | 19 | 12 | 31
  13 years | 17 | 23 | 40
  14 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 76 | 154
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 78 | 76 | 154
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 78 | 76 | 154
Language [Count of Participants; unit: Participants]
  English | 28 | 27 | 55
  Luganda | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received the Next HPV Vaccine Dose
Description: Timeliness of vaccination will be measured by the number of participants who received the next HPV vaccine dose.
Time Frame: Up to 6 months from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message Reminders | Usual Care
Number analyzed (Participants) | 78 | 76
Participants | 51 | 27

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Text Message Reminders | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/76
Other Adverse Events (participants affected / at risk) | 0/78 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT05151367/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05151367/SAP_001.pdf